CLINICAL TRIAL: NCT03302455
Title: A Randomized Controlled Study of E-aid Cognitive Behavior Therapy in Patients With Acute Insomnia to Prevent Transition to Chronic Insomnia
Brief Title: E-aid Cognitive Behavior Therapy for Insomnia to Prevent Transition From Acute Insomnia to Chronic Insomnia in China
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Nanfang Hospital, Southern Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: NFEC-2017-131
Record Dates: First submitted 2017-09-25; First posted 2017-10-05 (Actual); Last update posted 2020-10-20 (Actual); Status verified 2020-06

CONDITIONS: Insomnia
Keywords: insomia; eCBTI; internet; psychotherapy; guided self-help; psychological treatment
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: One group receives brief e-aid cognitive behavior therapy, and the other group does not receive any interventions during a clinical study.
Who Masked: Outcomes Assessor
Masking Description: The independent researcher from the IT department who carries out the randomisation and allocation procedure will be blinded to the study protocol. Participants could not be blinded to treatment allocation as participants in the control group did not receive any intervention from this trial. The research team will have limited contact with both IT staff and study participants, therefore, will not be able to bias the allocation or the assessments. Statistical analyses will be carried out by an independent researcher from the Southern Medical University who is not involved with the randomisation and assessment procedures.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- eCBTI (Experimental): This group will receive a 1-week of eCBTI treatment and will receive 3 months of follow-up.
  Interventions: Behavioral: eCBTI
- Control (No Intervention): This group does not receive any interventions during first 3 months of clinical study. If the participants still have no remission from insomnia after 3 months, will be recommended to enter the standardized insomnia treatment (medication and / or non-drug treatment).

INTERVENTIONS:
Behavioral: eCBTI — The brief eCBTI contains a one-week core course: sleep hygiene education, sleep restriction, stimulus control, relaxation audios, cognitive components, information about sleeping pills, and a brief overview. In addition, individual customized sleep restriction and stimulation control treatments were provided according to the subject's previous 2-week sleep status.
  Arms: eCBTI

SUMMARY:
Acute insomnia is one of the most common sleep disorders. Online cognitive behavioral therapy for insomnia (e-aid Cognitive Behavioral Therapy for Insomnia, eCBTI) has received wide attention in recent years. Foreign countries already have some eCBTI treatment tool, shown similar efficacy as standard CBTI, but how eCBTI can help in acute insomnia require further exploration and examination.

In this study, Investigators will establish eCBTI treatment tool to test whether eCBTI can reduce the conversion of acute insomnia to chronic insomnia disorder; and whether they can improve insomnia symptoms, sleep-related symptoms, anxiety and depressive symptoms, and quality of life

DETAILED DESCRIPTION:
Insomnia patients are collected from: Outpatients from Sleep clinics. Included 200 cases of acute insomnia patients, the participants will randomly divided into 100 brief eCBTI Group and 100 patients with control group, brief eCBTI Group will receive 1 Week eCBTI intervention and control group will not receive any intervention. Both groups will receive 3 months of follow-up.

At week 2, ISI and HADS will be conducted. Brief eCBTI group will also complete Treatment Component Adherence Scale (TCAS) in order to assess treatment adherence to and perceived helpfulness of each therapeutic element. At 3 months, two groups of subjects will have baseline assessment(except socio-demographic information), including chronic insomnia disorder diagnosis and self evaluation form (ISI, DBAS, SHPS ,PSAS,FIRST,ESS,HADS,SF-12v2).

This study provides a Smartphone to complete third-party applications online insomnia treatment procedures. Brief eCBTI includes 1-week core curriculum: sleep hygiene education, sleep restriction, stimulus control, relaxation audios, cognitive components, information about sleeping pills, and a brief overview.

Previous studies have shown that approximately 40% of acute insomnia will turn into Chronic insomnia disorder.While our preliminary work suggests, with the extension of follow-up time, high rates of chronic insomnia may be more ( 52.3% ).In order to meet the 95% confidence intervals (Confidence Interval, CI )( 35%-49% ) requirement, the project needs 200 acute insomnia disorder subjects, and random access eCBTI Treatment group and the control group (100 Cases) of whom an estimated 70% or more participants can complete 3 months of follow-up. This sample size ensures continuous data of small sample (Cohen d = 0.30) statistical effect is greater than 0.8, And test the odds ratio of dichotomous variables (Odds Ratio, OR) greater than 1.50(p>0.05 ).

Mean value for continuous variable data ± Standard deviation, Numerical or categorical variable data expressed as a percentage. T test for the continuous variables and Chi Square test for the categorical variables will be used. Using repeated measures analysis of variance to compare two sets of continuous variables in the treatment and follow-up of changes in the process (such as ISI score, etc). Incidence of chronic insomnia is computed using Chi Square test. All statistical procedures are used in Windows running 26.0 version of the SPSS package (IBM SPSS 26.0).

ELIGIBILITY:
Inclusion Criteria:

* Clinical diagnosis for acute insomnia according to the Diagnostic and Statistical Manual of Mental Disorders, Fifth Edition (DSM-5);
* Must be eighteen years or older;
* Must be able to comply with the intervention;
* Must be able to provide informed consent;
* Owning smart devices (such as smartphones and tablets).

Exclusion Criteria:

* A significant untreated mental or medical illness (e.g. consciousness disturbances, mania, acute phase of schizophrenia, major depressive disorder);
* Received any kind of psychological treatment for insomnia in the past 6 months;
* Shift workers, frequent cross-time flyers (e.g. shifted nurse/health professionals, international flight crew).

To allow for greater generalisability, this study does not exclude patients with a stable condition of somatic disease, mental disorders (eg, depression in remission), or individuals receiving pharmacological treatments (eg, antihypertensive drugs, antidepressants and benzodiazepines).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 192 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2019-06-02 (Actual); Study Completion 2019-06-02 (Actual)

PRIMARY OUTCOMES:
Incidence of chronic insomnia | 3 months
  the diagnostic criteria for chronic insomnia disorder according to DSM-5

SECONDARY OUTCOMES:
Changes in Ford Insomnia Response to Stress Test (FIRST) | baseline and 3 months
  FIRST, a measure to identify individuals predisposed to sleep disturbance and the subsequent development of chronic insomnia. This nine-item self-report instrument assesses the potential likelihood that an individual will experience sleep disturbance following various stressful events/situations. FIRST scores range from 9 to 36.
Changes in Short Form 12-Item Health Survey version 2（SF-12v2） | baseline and 3 months
  The SF-12v2 is a 12-item self-report questionnaire used to assess generic health outcomes from the patient's perspective.The SF-12v2 addresses the 8 domains viz. Physical functioning (PF), Role - physical (RP),Bodily pain (BP),General health perceptions (GH),Vitality (V),Social functioning (SF),Role - emotional (RE) and Mental health (MH) . The 2 scores that will be obtained from this assessment are composite scores representing physical health and mental health composite summaries, PCS and MCS respectively.
Changes in Sleep Hygiene and Practices Scale(SHPS) | baseline and 3 months
  Subjects' general sleep hygiene and practices are measured with Sleep Hygiene and Practices Scale.The SHPS is a 30-item self-report measure designed to assess the practice of sleep hygiene behaviors. Each item is rated on a six-point scale ranging from 1 to 6 . Total scores range from 30 to 180. SHPS has shown adequate reliability and validity .
Changes in Pre-Sleep Arousal Scale(PSAS) | baseline and 3 months
  Participant's problems during initiation of sleep is assessed with Pre-Sleep Arousal Scale.The Pre-Sleep Arousal Scale (PSAS) is a brief self-administered measure in which participants rate the intensity of experienced arousal. Internal consistency for somatic (8 items) and cognitive (8 items) subscales are satisfactory (α = 0.81 and α = 0.76) respectively.
Changes in Epworth Sleepiness Scale(ESS) | baseline and 3 months
  Subjective measure of a patient's sleepiness is measured with Epworth Sleepiness Scale.The Epworth Sleepiness Scale is a self-report 8-item questionnaire producing scores from 0 to 24. Scores greater than 10 suggest significant daytime sleepiness. The Epworth Sleepiness Scale has good psychometric properties , correlates with objective measures of sleepiness , and has been shown to differentiate between individuals with and without sleep disorders and those who are and are not sleep deprived.
Changes in Hospital Anxiety and Depression Scale (HADS) | baseline, week 2, and 3 months
  The HADS is a self-report questionnaire to determine the levels of anxiety and depression that a participant is experiencing. The HADS is a fourteen item scale that generates ordinal data. Seven of the items relate to anxiety and seven relate to depression.Each item on the questionnaire is scored from 0-3 and this means that a person can score between 0 and 21 for either anxiety or depression. For anxiety (HADS-A) this gave a specificity of 0.78 and a sensitivity of 0.9. For depression (HADS-D) this gave a specificity of 0.79 and a sensitivity of 0.83.
Treatment Component Adherence Scale (TCAS) | week 2
  A self-reported questionnaire will be administered posttreatment to assess adherence to CBTI guidelines and the perceived helpfulness of treatment guidelines. Adherence to each therapeutic element will be rated on a 0 to 3 scale as follows: (0) Followed rarely or not at all; (1) Followed occasionally; (2) Followed most of the time; (3) Followed consistently. Ratings for all therapeutic elements will be broadly grouped into a Behavioral Component and a Cognitive Component.
Changes in Dysfunctional Beliefs and Attitudes about Sleep Scale (DBAS) | baseline and 3 months
  The DBAS is a 30-item self-report questionnaire designed to evaluates sleep-related beliefs, querying respondents' expectations and attitudes regarding the causes, consequences, and potential treatments of sleep issues. The 30-item version showed adequate psychometric properties as evidenced by good internal consistency (Cronbach Alpha = 0.80), moderate item-total correlations (mean rs = 0.37), and adequate convergent and discriminant validity.Likert-type scale requiring participants to choose from 1 to 5 will be used. Thus, the results are quantified in terms of strength of endorsed beliefs. A higher score indicates more dysfunctional beliefs and attitudes about sleep. The total score is based on the average score of all items.
Changes in Insomnia Severity Index(ISI) | baseline，week 2, and 3 months
  The ISI is a 7-item self-report questionnaire assessing the nature, severity, and impact of insomnia in the last month. The dimensions evaluated are: severity of sleep onset, sleep maintenance, and early morning awakening problems, sleep dissatisfaction, interference of sleep difficulties with daytime functioning, noticeability of sleep problems by others, and distress caused by the sleep difficulties. A 5-point Likert scale is used to rate each item (e.g., 0 = no problem; 4 = very severe problem), yielding a total score ranging from 0 to 28.

CONTACTS AND LOCATIONS:
Overall Officials: Bin Zhang, MD & PhD, Principal Investigator — Nanfang Hospital, Southern Medical University
Locations (1):
- Nanfang Hospital, Southern Medical University, Guangzhou, Guangdong, China

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Yang Y, Luo X, Paudel D, Zhang J, Li SX, Zhang B. Effects of e-aid cognitive behavioural therapy for insomnia (eCBTI) to prevent the transition from acute insomnia to chronic insomnia: study protocol for a randomised controlled trial. BMJ Open. 2019 Nov 18;9(11):e033457. doi: 10.1136/bmjopen-2019-033457. PMID 31740476